CLINICAL TRIAL: NCT06736535
Title: Prevalence of Hypomineralized Second Primary Molars and Its Association With Hypomineralized Primary Canines In A Group of Egyptian Children: A Cross-Sectional Study.
Brief Title: Prevalence of Hypomineralized Second Primary Molars In A Group of Egyptian Children
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Farida Khalid Noaman, Prevalence of Hypomineralized Second Primary Molars and Its Association with Hypomineralized Primary Canines In A Group of Egyptian Children, Cairo University
Other Study IDs: HPC in Egyptian Children
Record Dates: First submitted 2024-12-12; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Hypomineralization of Enamel
MeSH Terms: conditions — Dental Enamel Hypomineralization

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim of the study: This study aims to detect the prevalence of hypomineralized second primary molars and its association with hypomineralized primary canines in a group of Egyptian children. Furthermore, it also addresses the possible etiological factors that might predispose hypomineralization of deciduous teeth.

Rationale:

This study tends to fill the knowledge gap about the prevalence of hypomineralized second primary molars as well as its association with hypomineralized primary canines in a group of Egyptian children. In addition to identifying the possible predisposing etiological factors.

DETAILED DESCRIPTION:
Developmental defects of enamel are common among deciduous and permanent dentition. One of these defects is termed molar incisor hypomineralization which refers to a qualitative defect in the enamel due to disruption in the process of calcification and maturation of ameloblasts. The most remarkable clinical appearance of the lesion is the weak quality of enamel which leads to teeth being susceptible to decay .

In 2011 a standardized scoring criteria was introduced by the European Academy of Pediatric Dentistry for proper diagnosis of MIH. Moreover, to distinguish MIH from other developmental enamel defects. Due to the poor quality of enamel, patients with MIH are prone to several challenges like hypersensitivity, dental pain and post eruptive enamel breakdown which creates drawbacks for the dentist to properly manage the case

A study conducted in 2013 referred to MIH occurring in primary dentition and was primarily termed as deciduous molar hypomineralization (DMH). Teeth was recorded using EAPD diagnostic criteria and the prevalence of DMH was 4% in teeth examined in a sample of 6,487 participating children. In addition, they found that the occurrence of MIH in children affected with HSPM was of higher results. Furthermore, children with more than one affected molar represented severe form of HSPM.

Another study conducted on Iraqi children to detect the prevalence and severity of HSPM on a sample of 809 children aging 7-9 years showed 6.6%. By using the EAPD scoring criteria and International Caries Detection and Assessment System the study revealed that more severe form of caries was proportional with the amount of demarcated lesion, moreover 39.6% of the cases examined showed correlation between HSPM and MIH.

The American Academy of Pediatric Dentistry in 2017 published a study that detected the prevalence of HSPM and HPC in a group of 1963 schoolchildren, the results were 6.48% and 2.22% respectively by adapting the EAPD scoring criteria and the Caries Assessment Spectrum and Treatment. Considering the severity, 70% of the affected cases reported mild to moderate hypomineralization. Furthermore, the study reported children diagnosed with HSPM or HPC are six times more likely to develop MIH.

Another study was implemented in 2021 to detect prevalence of HSPM/HPC and to mark out the lesion characteristics, location and severity. Guided by the EAPD scoring criteria the results are as follows, in a sample of 153 patients HSPM showed 18.95% and HPC showed 11.11%. The lesions were mostly detected on the buccal and occlusal surfaces. This study measured the severity in 153 samples to report majority of lesions exhibiting mild degree severity.

A study that was conducted in North India to detect the prevalence of HSPM showed 7.9% in a sample of 300 patients. In addition to determining the possible etiological factors behind the occurrence of HSPM. The etiology remains uncertain, however based on the data collected from medical reports and from the parents, the study concluded that prenatal and post-natal factors showed higher prevalence of HSPM than perinatal factors.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4-9 years.
* Cooperative patients.
* Medically Free children.
* Both Genders; females and males will be included.

Exclusion Criteria:

* Non-Egyptian nationality.
* Special Health Care Needs Patients.
* Other developmental enamel defects (Non-MIH/HSPM); Amelogenesis Imperfecta, dental fluorosis and hypoplasia.
* Other medical syndromes.

Ages: 4 Years to 9 Years | Sex: All
Age Groups: Child
Study Population: Children attending Outpatient clinics of Cairo University will be recruited in the study.
Sampling Method: Non-Probability Sample
Enrollment: 825 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of HPC in Egyptian Children | Baseline
Prevalence of HSPM in Egyptian Children | Baseline

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bekes K, Steffen R, Kramer N. Hypomineralised second primary molars: the Wurzburg concept. Eur Arch Paediatr Dent. 2024 Aug;25(4):597-602. doi: 10.1007/s40368-024-00913-7. Epub 2024 May 28. PMID 38805129
- [Background] da Silva Figueiredo Se MJ, Ribeiro APD, Dos Santos-Pinto LAM, de Cassia Loiola Cordeiro R, Cabral RN, Leal SC. Are Hypomineralized Primary Molars and Canines Associated with Molar-Incisor Hypomineralization? Pediatr Dent. 2017 Nov 1;39(7):445-449. PMID 29335050
- [Background] Elfrink ME, Ghanim A, Manton DJ, Weerheijm KL. Standardised studies on Molar Incisor Hypomineralisation (MIH) and Hypomineralised Second Primary Molars (HSPM): a need. Eur Arch Paediatr Dent. 2015 Jun;16(3):247-55. doi: 10.1007/s40368-015-0179-7. Epub 2015 Apr 18. PMID 25894247
- [Background] Borrego-Marti N, Peris-Corominas R, Maura-Solivellas I, Ferres-Padro E, Ferres-Amat E. Hypomineralisation of second primary molars and primary canines: Prevalence and description of lesions in a population of 153 patients visited at a hospital paediatric dentistry service. Eur J Paediatr Dent. 2021 Sep;22(3):237-242. doi: 10.23804/ejpd.2021.22.03.11. PMID 34544254
- [Background] Lygidakis NA, Garot E, Somani C, Taylor GD, Rouas P, Wong FSL. Best clinical practice guidance for clinicians dealing with children presenting with molar-incisor-hypomineralisation (MIH): an updated European Academy of Paediatric Dentistry policy document. Eur Arch Paediatr Dent. 2022 Feb;23(1):3-21. doi: 10.1007/s40368-021-00668-5. Epub 2021 Oct 20. PMID 34669177